CLINICAL TRIAL: NCT00670345
Title: Efficacy of Tranexamic Acid in Reducing Perioperative Bleeding in Patients Undergoing Radical Prostatectomy. A Randomized Controlled Double-blind Study.
Brief Title: Tranexamic Acid in Urologic Surgery
Acronym: TRANEX-URO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GO/URC/ER/mm 139/DG
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2010-07

CONDITIONS: Bleeding; Prostatectomy
Keywords: tranexamic acid; prostatectomy; surgery
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Patients will receive a slow endovenous infusion of 500 mg of tranexamic acid before surgical incision, followed by 250 mg/h of tranexamic acid by continuous infusion.
  Interventions: Drug: Tranexamic Acid
- 2 (Placebo Comparator): Patients belonging to the control group will receive the same volume of saline infusions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Patients will receive a slow endovenous infusion of 500 mg of tranexamic acid before surgical incision, followed by 250 mg/h of tranexamic acid by continuous infusion.
  Other Names: TRANEX; UGUROL
  Arms: 1
Drug: Placebo — Patients belonging to the control group will receive the same volume of saline infusions.
  Arms: 2

SUMMARY:
This prospective randomized double-blind placebo vs control study aims at verifying the efficacy of tranexamic acid administration in reducing perioperative bleeding in patients undergoing open radical prostatectomy. Two recent meta-analysis confirmed that tranexamic acid administration does not increase mortality, myocardial infarction, deep venous thrombosis, pulmonary embolism, stroke and renal failure.

200 patients undergoing open radical prostatectomy will be enrolled. Patients will receive a slow endovenous infusion of 500 mg of tranexamic acid before surgical incision, followed by 250 mg/h of tranexamic acid by continuous infusion.

Patients belonging to the control group will receive the same volume of saline infusions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients undergoing open radical prostatectomy

Exclusion Criteria:

* Age < 18 years
* Patients with drug eluting stent with a double antiplatelet therapy
* Atrial fibrillation
* Thrombophilic diathesis
* Allergy to tranexamic acid

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-04; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Landoni, MD, Study Director — Università Vita-Salute San Raffaele, Milano, Italia e Istituto Scientifico San Raffaele, Milano, Italia; Antonella Crescenti, MD, Principal Investigator — Università Vita-Salute San Raffaele, Milano, Italia e Istituto Scientifico San Raffaele, Milano, Italia
Locations (1):
- Università Vita-Salute San Raffaele, Milano, Italia e Istituto Scientifico San Raffaele, Milano, Italia, Milan, Italy

REFERENCES:
- [Result] Crescenti A, Borghi G, Bignami E, Bertarelli G, Landoni G, Casiraghi GM, Briganti A, Montorsi F, Rigatti P, Zangrillo A. Intraoperative use of tranexamic acid to reduce transfusion rate in patients undergoing radical retropubic prostatectomy: double blind, randomised, placebo controlled trial. BMJ. 2011 Oct 19;343:d5701. doi: 10.1136/bmj.d5701. PMID 22012809